CLINICAL TRIAL: NCT05571839
Title: A Phase 1 Study of PF-08046049/SGN-BB228 in Advanced Melanoma and Other Solid Tumors
Brief Title: A Study of PF-08046049/SGN-BB228 in Advanced Melanoma and Other Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGNBB228-001; C5871001 (Other: Alias Study Number); 2022-502348-11-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Cutaneous Melanoma; Non-small Cell Lung Cancer; Colorectal Neoplasms; Pancreatic Neoplasms; Mesothelioma
Keywords: NSCLC; Colorectal Cancer; CRC; Pancreatic Cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Pancreatic Neoplasms; Mesothelioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-08046049 (Experimental): PF-08046049 monotherapy
  Interventions: Drug: PF-08046049

INTERVENTIONS:
Drug: PF-08046049 — Given into the vein (IV; intravenous)

SUMMARY:
This study will test the safety of a drug called PF-08046049/SGN-BB228 in participants with melanoma and other solid tumors that are hard to treat or have spread through the body. It will also study the side effects of this drug. A side effect is anything a drug does to the body besides treating the disease.

This study will have 3 parts. Parts A and B of the study will find out how much PF-08046049/SGN-BB228 should be given to participants. Part C will use the information from Parts A and B to see if PF-08046049/SGN-BB228 is safe and if it works to treat solid tumor cancers.

ELIGIBILITY:
Inclusion Criteria:

* All Parts: Participants must have disease that is relapsed, refractory, or intolerant to standard of care. Participants must have histologically or cytologically confirmed metastatic malignancy.
* Participants must have one of the following tumor types:

  * Parts A and B: Participants must have metastatic or unresectable cutaneous melanoma.
  * Part C: Participants must have one of the following tumor types:

    * Cutaneous Melanoma
    * Non-small Cell Lung Cancer (NSCLC)
    * Colorectal Cancer (CRC)
    * Pancreatic Cancer
    * Mesothelioma
* A pre-treatment biopsy or submission of archival tissue is required
* For participants with cutaneous melanoma

  * Must have been previously treated with an anti-programmed death-1 (anti-PD-1) or anti-programmed death ligand-1 (anti-PD-L1) agent given alone or with other therapies.
  * Participants with a targetable BRAF mutation must have been treated with, been intolerant of, or been deemed ineligible to receive treatment with BRAF/MEK targeted therapy prior to study entry.
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
* Measurable disease per RECIST v1.1 at baseline

Exclusion Criteria:

* History of another malignancy within 3 years before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy. Exceptions are malignancies with a negligible risk of metastasis or death.
* Active central nervous system metastases or leptomeningeal disease. Participants with previously treated brain metastases may participate provided they are:

  * clinically stable for at least 4 weeks prior to study entry after brain metastasis treatment,
  * they have no new or enlarging brain metastases,
  * and are off of corticosteroids prescribed for symptoms associated with brain metastases for at least 7 days prior to the first dose of study drug.
* Prior therapies cannot include any drugs targeting CD228 or 4-1BB
* Immunotherapy, biologics, and/or other approved or investigational antitumor treatment that is not completed 4 weeks prior to first dose of study drug, or within 2 weeks prior to the first dose of study drug if the underlying disease has progressed on treatment
* Melanoma subtypes including acral, uveal, and mucosal are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2026-06-06 (Estimated); Study Completion 2026-06-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Through 30 days after the last study treatment; approximately 7 months
  Any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Number of participants with laboratory abnormalities | Through 30 days after the last study treatment; approximately 7 months
Number of participants with dose limiting toxicities | Up to 28 days

SECONDARY OUTCOMES:
Number of participants with antidrug antibodies | Through 30 days after the last study treatment; approximately 7 months
  To be summarized using descriptive statistics
Pharmacokinetic (PK) parameter - Area under the curve (AUC) | Through 30 days after the last study treatment; approximately 7 months
  To be summarized using descriptive statistics
PK parameter - Maximum Concentration (Cmax) | Through 30 days after the last study treatment; approximately 7 months
  To be summarized using descriptive statistics
PK parameter - Time to maximum concentration (Tmax) | Through 30 days after the last study treatment; approximately 7 months
  To be summarized using descriptive statistics
PK parameter - Apparent terminal half-life (t1/2) | Through 30 days after the last study treatment; approximately 7 months
  To be summarized using descriptive statistics
PK parameter - Trough concentration (Ctrough) | Through 30 days after the last study treatment; approximately 7 months
  To be summarized using descriptive statistics
Objective response rate (ORR) | Up to approximately 1 year
  The proportion of participants with a complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as assessed by the investigator
Duration of response (DOR) | Up to approximately 1 year
  The time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of progressive disease (PD) (based on radiographic assessments per RECIST v1.1) or death due to any cause
Progression-free survival (PFS) | Up to approximately 1 year
  The time from the start of study treatment to the first documentation of PD (per RECIST v1.1 as assessed by the investigator) or death due to any cause
Overall survival (OS) | Approximately 2 years
  The time from the start of study treatment to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (35):
- United States (27):
  - UCLA Hematology/Oncology - Administrative Office, Los Angeles, California
  - The Angeles Clinic and Research Institue, A Cedars-Sinai Affiliate, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Drug Information Center, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - UCLA Hematology/ Oncology- Pasadena, Pasadena, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - UCSF Medical Center, Investigational Pharmacy, San Francisco, California
  - UCLA Hematology/Oncology - Santa Barbara, Santa Barbara, California
  - The Angeles Clinic and Research Institute, A Cedars-Sinai Affiliate (Emergency Back-up only), Santa Monica, California
  - UCLA Hematology - Oncology Clinic - Westlake Village, Westlake Village, California
  - Quest Diagnostics Incorporated - Denver, Denver, Colorado
  - Presbyterian/St. Lukes Medical Center, Denver, Colorado
  - Northwestern Medical Group, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - BWH, Boston, Massachusetts
  - Dana-Farber Cancer Institute (DFCI), Boston, Massachusetts
  - Laboratory Corporation of America, Raritan, New Jersey
  - Ambulatory Care Center at NYU Langone Medical Center, New York, New York
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - NYU Langone Hospitals, NYU Langone Rusk Ambulatory Surgical Pharmacy, New York, New York
  - NYU Langone Medical Center(Tisch Hospital), New York, New York
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Baylor Sammons Cancer Center, Dallas, Texas
  - US Oncology Investigational Products Center (IPC), Irving, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Canada (3):
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- France (2):
  - Insitut Gustave Roussy, Villejuif, Cedex
  - Institut Gustave Roussy, Villejuif
- Clinical Research Center Dermatology (CRCD) Dermatoonkologie Charité - Universitätsmedizin Berlin, Berlin, Germany
- UniversitätsSpital Zürich Dermatologische Klinik, Zurich, Switzerland
- The Beatson West of Scotland Cancer Centre, Glasgow, Glasglow CITY, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGNBB228-001